CLINICAL TRIAL: NCT06665542
Title: A Multicenter Prospective Observational Study to Derive and Verify the Performance of a Host-response Based Diagnostic Tool for Early Detection of Severe Infections.
Status: Active, not recruiting | Type: Observational
Sponsor: MeMed Diagnostics Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: MMD01SEV
Record Dates: First submitted 2024-10-28; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Sepsis; Acute Infection
Keywords: Host response; Suspected sepsis; Suspected acute infection; Biomarkers; ARDS; Septic shock; Sepsis associated AKI
MeSH Terms: conditions — Sepsis; Shock, Septic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples Without DNA — Plasma , Serum , whole Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Suspected infection/sepsis: Patient presenting with a clinical suspicion of acute infection/sepsis as defined by the attending physician, based on clinical presentation.
- Healthy Individuals: No clinical suspicion of acute infection.

SUMMARY:
The study is a multi-center, prospective, observational clinical study enrolling patients from at least 3 medical centers. Study population will include patients over the age of 18 years.

The study will recruit patients presenting with suspicion of acute infection/sepsis and healthy individuals.

Study main objective is to derive and verify a host response based score to predicte severe outcome.

DETAILED DESCRIPTION:
For determining disease severity each enrolled patient will be assigned as either "severe outcome patient" or "non severe outcome patient" according to predefined criteria. (or "healthy").

Participation in the study requires the collection of routine patient data and blood sample. Blood samples will be used for measurements of host biomarkers that predict disease severity. The blood samples will be collected upon enrollment.

In addition, a standardized patient questionnaire inquiring about severity outcomes met up to 28 days after presentation will be conducted by phone call 28 to 42 days post admission.

Enrolled patients will be managed according to the current standard of care per standard institutional procedures. Results of the measured biomarkers will not be revealed to the attending clinician and so will not influence patient management.

ELIGIBILITY:
Suspected acute infection/sepsis patients

Patients eligible for inclusion are required to fulfill all of the following criteria:

* Written informed consent must be obtained from the patient or his/her legal guardian.
* Over 18 years of age
* Clinical suspicion of acute infection/sepsis as defined by the attending physician, based on clinical presentation.

Healthy individuals

Patients eligible for inclusion are required to fulfill all of the following criteria:

* Written informed consent must be obtained from the patient
* Over 18 years of age
* No clinical suspicion of acute infection.

Exclusion Criteria:

Suspected acute infection/sepsis patients

Patients fulfilling the following criteria are not eligible for inclusion in this study:

* HIV, HBV, active HCV or active Tuberculosis infection (self-declared or known from medical records).
* Pregnancy- self reported or medically confirmed. Healthy individuals

Patients fulfilling the following criteria are not eligible for inclusion in this study:

* Episode of infection in the last 2 weeks
* Major trauma and\or burns and\or surgery in the last 2 weeks
* HIV, HBV, active HCV or active Tuberculosis infection (self-declared or known from medical records)
* Elective surgery patients
* Pregnancy- self reported or medically confirmed

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patients presenting with suspected infection/sepsis as defined by the attending physician, based on clinical presentation and laboratory/radiological findings. Additionally, the study will recruit healthy individuals across all study sites.
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2020-11-12 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary objective | 3,14 and 28 Days
  To derive and verify the diagnostic performance of a host-response tool based on novel biomarkers for predicting disease severity in adult patients, aged 18 years or older, presenting with clinical suspicion of acute infection/sepsis.

CONTACTS AND LOCATIONS:
Locations (8):
- United States (2):
  - Maimonides MC, New York, New York
  - MCW, Milwaukee, Wisconsin
- Israel (6):
  - Carmel MC, Haifa
  - Rambam MC, Haifa
  - Edith Wolfson MC, Holon
  - Shaare Zedek MC, Jerusalem
  - Beilinson MC, Petah Tikva
  - Sheba Tel-HaShomer MC, Tel Aviv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC6015097/
- See also: Related Info — https://www.researchgate.net/publication/324702741_Evaluation_of_Antibiotics_Prescriptions_in_the_City_of_Vitoria_ES_-_Brazil_and_its_Relation_with_Laboratory_Diagnosis
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC9484674/
- See also: Related Info — https://pmc.ncbi.nlm.nih.gov/articles/PMC3159846/
- See also: Related Info — https://www.researchgate.net/publication/23177948_Role_of_the_eosinophil_count_in_discriminating_the_severity_of_community-acquired_pneumonia_in_HIV-infected_patients
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/28114554/
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/31583025/
- See also: Related Info — https://www.researchgate.net/publication/331851658_Combining_quick_sequential_organ_failure_assessment_score_with_heart_rate_variability_may_improve_predictive_ability_for_mortality_in_septic_patients_at_the_emergency_department
- See also: Related Info — https://bmjopen.bmj.com/content/6/9/e011021